CLINICAL TRIAL: NCT03954444
Title: A Randomized, Double Blind, Parallel Group, Three Arm, Placebo Controlled, Multi-Site Therapeutic Equivalence Study With Clinical End-points Comparing Test Product "Oxymetazoline Hydrochloride Cream, 1%" to Reference Product "RHOFADETM Cream, 1%" in the Treatment of Moderate to Severe Persistent Facial Erythema of Rosacea
Brief Title: A Clinical Endpoint Bioequivalence Study of "Oxymetazoline Hydrochloride Cream"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXY2018-01
Record Dates: First submitted 2019-04-10; First posted 2019-05-17 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oxymetazoline hydrochloride Cream, 1% (Active Comparator): Oxymetazoline hydrochloride cream, 1%
  Interventions: Drug: Oxymetazoline Hydrochloride
- RHOFADE Cream, 1% (Active Comparator): RHOFADE Cream, 1%
  Interventions: Drug: Rhofade Cream, 1%
- Vehicle Cream (Placebo Comparator): Vehicle cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxymetazoline Hydrochloride — Test Comparator
  Arms: Oxymetazoline hydrochloride Cream, 1%
Drug: Rhofade Cream, 1% — Reference Comparator
  Other Names: Oxymetazoline hydrochloride
  Arms: RHOFADE Cream, 1%
Drug: Placebo — Placebo Comparator
  Other Names: Oxymetazoline hydrochloride
  Arms: Vehicle Cream

SUMMARY:
A Randomized, Double-blind, Parallel-group, Three-arm, Placebo-controlled, Multi-Site Therapeutic Equivalence Study with Clinical End-points Comparing Test Product "Oxymetazoline hydrochloride Cream, 1%" to Reference Product "RHOFADE™ Cream, 1%" in the Treatment of Moderate to Severe Persistent Facial Erythema of Rosacea

ELIGIBILITY:
Inclusion Criteria:

* (1) Study subjects must have provided IRB approved written informed consent using the latest version of the IRB informed consent form, (or assent in applicable states/countries). In addition, study subjects must sign a HIPAA authorization, if applicable.
* (2) Healthy male or non-pregnant females, ≥18 years-of-age with a clinical diagnosis of rosacea with persistent (non-transient) facial erythema.
* (3) Ability to follow study instructions and complete subject diary without assistance.
* (4) Females of child bearing potential must not be pregnant or lactating at screening visit and at baseline visit, as documented by a negative urine pregnancy test.
* (5) Female subjects of childbearing potential must be willing to use an acceptable form of birth control from the day of the first dose administration to 30 days after the last administration of Investigational Product (IP). A sterile sexual partner is NOT considered an adequate form of birth control.
* (6) Moderate to severe persistent facial erythema associated with rosacea, defined as a grade of ≥3 on the CEA scale as assessed by the Investigator at Screening and on Baseline (Day 1) visit prior to study drug application.
* (7) Moderate to severe persistent facial erythema associated with rosacea, defined as a grade of ≥3 on the SSA scale as assessed by the subject at Screening and on Baseline (Day 1) visit prior to study drug application.
* (8) Stable erythema (for at least 3 months prior to screening) associated with rosacea, with minimal variation from day to day and within each day, in the opinion of the subject.
* (9) Willingness to complete the required visits including short stay for at least 12 hours at the investigational site for 2 separate visits.
* (10) Subjects who use make-up, facial moisturizers, creams, lotions, cleansers and/or sunscreens must have used the same product brands/types for a minimum period of 4 weeks prior to Baseline, must agree not to change brand/type or frequency of use throughout the study and must agree not to use make-up, facial moisturizers, creams, lotions and/or sunscreens on the scheduled clinic visit day before the visit.
* (11) Subject must be willing to avoid the use of abrasive cleansers or washes (e.g., exfoliating facial scrubs), adhesive cleansing strips (e.g., Bioré® Pore Strips) and wax epilation on the face, during the entire duration of their study participation.
* (12) Subject's willingness to minimize external factors that might trigger rosacea flare-ups (e.g., spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds, alcoholic beverages).
* (13) Subject must be in good health and free from any systemic or dermatological disorder (other than rosacea) that, in the opinion of the Investigator, will interfere with the study evaluations or increase the risk of AEs.
* (14) Any skin type or race, providing the skin pigmentation will allow discernment of erythema.

Exclusion Criteria:

* (1) Any of the following conditions: severe or unstable or uncontrolled cardiovascular disease, clinically unstable hypertension, orthostatic hypotension, and uncontrolled hypertension or hypotension, cerebral or coronary insufficiency, Raynaud's Syndrome, thromboangiitis obliterans, scleroderma, Sjögren's syndrome, renal or hepatic impairment.
* (2) Subjects with narrow angle glaucoma.
* (3) Females who are pregnant, breast feeding, or planning a pregnancy during the study.
* (4) Females of childbearing potential who do not agree to utilize an adequate form of contraception during their participation in the study.
* (5) Clinical signs of particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) on the face or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia that may interfere with the study evaluations, in the opinion of the Investigator.
* (6) Presence of ≥3 facial inflammatory lesions of rosacea at screening and baseline.
* (7) Presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea, as determined by the Investigator.
* (8) Excessive facial hair (e.g., beards, sideburns, moustaches, etc.) that would interfere with the study treatments or study assessments.
* (9) History of drug or alcohol abuse within 12 months prior to the Screening visit.
* (10 Known hypersensitivity or allergies to any component of the study treatment.
* (11) Use within 12 hours prior to baseline of any topical products including, but not limited to, lotions, creams, ointments, and cosmetics applied to the face (facial cleanser is acceptable).
* (12) Use 1 week prior to baseline of niacin ≥500 mg/day.
* (13) Use within 2 weeks prior to baseline of products containing topical corticosteroids, topical retinoids, topical antibiotics, topical anti-inflammatory, topical treatment for rosacea, or topical treatment for acne.
* (14) Use within 4 weeks prior to baseline of topical immunomodulators, systemic antibiotics, systemic corticosteroids, systemic anti-inflammatory agents, systemic treatment for rosacea, or systemic treatment for acne (other than oral retinoids, which require a 6-month washout).
* (15) Undergone 4 weeks prior to baseline any dermatologic or surgical procedure on the face.
* (16) Use within 3 months prior to baseline of any systemic immunomodulators known to have an effect on rosacea.
* (17) Use within 6 months prior to baseline of any oral retinoids (e.g., isotretinoin) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* (18) Undergone 6 months prior to baseline any laser, light-source (e.g. intense pulsed light, photodynamic therapy) or other energy-based therapy to the face.
* (19) Exposed to excessive UV radiation within 1 week before Screening visit and/or subject is unwilling to refrain from excessive exposure to UV radiation during the course of the study.
* (20) Current use of monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, alpha-agonists, cardiac glycosides, beta blockers, other antihypertensive agents, or oxymetazoline (e.g., eye drops, nasal sprays).
* (21) Subject has participated in a clinical trial within 30 days or in a biologics study within 6 months preceding admission of this study.
* (22) Previous participation in this study.
* (23) Inability to communicate well (i.e., language problem, poor mental development, psychiatric illness or poor cerebral function), that may impair the ability to provide written informed consent.
* (24) Subject has any evidence of organ dysfunction, chronic infectious disease, system disorder or has a condition or is in a situation that, in the Investigator's opinion, that may put the subject at significant risk, may confound the study results, or may significantly interferes with the subject's participation in the study.
* (25) Employees or family members of the research center or Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Lynchburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymetazoline Hydrochloride Cream, 1%: Oxymetazoline hydrochloride cream, 1%
  Oxymetazoline Hydrochloride: Test Comparator
  Subjects applied once daily to face for 29 days
- RHOFADE Cream, 1%: RHOFADE Cream, 1%
  Rhofade Cream, 1%: Reference Comparator
  Subjects applied once daily to face for 29 days
- Vehicle Cream: Vehicle cream
  Placebo: Placebo Comparator
  Subjects applied once daily to face for 29 days
Period: Overall Study
Arm/Group | Oxymetazoline Hydrochloride Cream, 1% | RHOFADE Cream, 1% | Vehicle Cream
Started | 379 | 382 | 344
Completed | 366 | 366 | 327
Not Completed | 13 | 16 | 17
Not completed — Withdrawal by Subject | 5 | 5 | 5
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Protocol Violation | 0 | 3 | 5
Not completed — Use of prohibited therapy | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Non-compliant with study drug application | 2 | 2 | 0
Not completed — Administrative reasons | 0 | 0 | 1
Not completed — Miscellaneous | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population also defined as in the Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxymetazoline Hydrochloride Cream, 1% | RHOFADE Cream, 1% | Vehicle Cream | Total
Number analyzed (Participants) | 379 | 382 | 344 | 1105
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (13.87) | 46.2 (14.01) | 47.2 (14.50) | 46.8 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 284 | 258 | 824
  Male | 97 | 98 | 86 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 202 | 205 | 182 | 589
  Not Hispanic or Latino | 177 | 177 | 162 | 516
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 9 | 2 | 4 | 15
  White | 369 | 377 | 337 | 1083
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Clinical Erythema Assessment Score [Count of Participants; unit: Participants]
  0-Clear | 0 | 0 | 0 | 0
  1-Almost Clear | 0 | 0 | 0 | 0
  2-Mild | 0 | 0 | 0 | 0
  3-Moderate | 287 | 292 | 273 | 852
  4-Severe | 92 | 90 | 71 | 253
Baseline Subject Self-Assessment [Count of Participants; unit: Participants] — Assessment of the severity of Rosacea at baseline.
  Subjects were graded on a scale from 0 = no rosacea to 4 = very severe rosacea
  Participants
    0-No Sign | 0 | 0 | 0 | 0
    1-Almost Clear | 0 | 0 | 0 | 0
    2-Mild | 0 | 0 | 0 | 0
    3-Moderate | 282 | 287 | 261 | 830
    4-Severe | 97 | 95 | 83 | 275

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment Success at All Time Points 3, 6, 9 and 12 Hours Post-application on Day 29. Treatment Success Was Defined as Having a Clinician Erythema Assessment Score at Least 2 Grades Lower Than the Baseline (Day 1 Predose) Value
Description: The primary efficacy endpoint was the proportion of subjects with treatment success at all time points 3, 6, 9, and 12 hours post-application on Day 29. Treatment success was defined as having CEA score at least 2 grades lower than the baseline (Day 1 pre-dose) value. Clinician Erythema Assessment was measured as (0-clear, 1-almost clear, 2-mild, 3-moderate, 4- severe).
Time Frame: 29 days
Population: Equivalence Analysis of the Primary Endpoint (Per Protocol Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxymetazoline Hydrochloride Cream, 1% | RHOFADE Cream, 1% | Vehicle Cream
Number analyzed (Participants) | 349 | 356 | 316
Participants
  Success | 78 | 70 | 51
  Failure | 271 | 286 | 265
Statistical Analysis 1: Comparison: Oxymetazoline Hydrochloride Cream, 1% vs RHOFADE Cream, 1%; Test type: Equivalence — 90% Confidence Interval, should be within -20% to +20%; Mean Difference (Net) = 2.7, 90% CI 2-sided [-2.6 to 8.0]
Statistical Analysis 2: Comparison: Oxymetazoline Hydrochloride Cream, 1% vs Vehicle Cream; Test type: Superiority; p = 0.04, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: RHOFADE Cream, 1% vs Vehicle Cream; Test type: Superiority; p = 0.1126, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 2 month adverse event data collection
Arm/Group | Oxymetazoline Hydrochloride Cream, 1% | RHOFADE Cream, 1% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/379 | 0/382 | 0/344
Serious Adverse Events (participants affected / at risk) | 0/379 | 1/382 | 1/344
Other Adverse Events (participants affected / at risk) | 61/379 | 60/382 | 48/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxymetazoline Hydrochloride Cream, 1% (N=379) | RHOFADE Cream, 1% (N=382) | Vehicle Cream (N=344)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxymetazoline Hydrochloride Cream, 1% (N=379) | RHOFADE Cream, 1% (N=382) | Vehicle Cream (N=344)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Androgen deficiency (Endocrine disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Application site acne (General disorders) | 4 | 6 | 2
Application site dermatitis (General disorders) | 3 | 2 | 1
Application site dryness (General disorders) | 5 | 2 | 1
Application site erythema (General disorders) | 7 | 10 | 7
Application site exfoliation (General disorders) | 0 | 0 | 1
Application site hypoaesthesia (General disorders) | 1 | 1 | 0
Application site irritation (General disorders) | 2 | 0 | 0
Application site pain (General disorders) | 9 | 16 | 10
Application site papules (General disorders) | 0 | 1 | 0
Application site paraesthesis (General disorders) | 1 | 0 | 0
Application site pruritus (General disorders) | 14 | 16 | 7
Application site rash (General disorders) | 2 | 0 | 0
Application site reaction (General disorders) | 8 | 2 | 1
Application site swelling (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Application site pustules (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 11 | 12
Migraine (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03954444/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03954444/SAP_001.pdf